CLINICAL TRIAL: NCT01080456
Title: A Randomized, Single Dose, Open Label, Bioequivalence Study of Tacrolimus Capsules 1 mg in Normal Healthy Male Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Tacrolimus 1 mg Capsule Under Fasting Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panacea Biotec Ltd (Industry)
Responsible Party: Dr. Arani Chatterjee, Panacea Biotec Ltd.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: US/07/052
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteers
Keywords: Bioequivalence study in healthy volunteers
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prograf® Capsule 1 mg (Active Comparator)
  Interventions: Drug: Tacrolimus 1 mg capsule
- Tacrolimus Capsule 1 mg (Experimental)
  Interventions: Drug: Tacrolimus 1 mg capsule

INTERVENTIONS:
Drug: Tacrolimus 1 mg capsule — Subjects will be administered either Test Product or Reference Product with 240 mL of water according to randomization schedule
  Other Names: Tacrolimus Capsule

SUMMARY:
The objective of the study is to demonstrate bioequivalence between Test Product (A): Tacrolimus Capsules 1 mg, manufactured by Panacea Biotec Limited, India and the corresponding Reference Product (B): Prograf (Tacrolimus) Capsules 1 mg, manufactured by Astellas Pharma, Inc., USA in 36 normal, healthy, adult, male subjects under fasting condition.

DETAILED DESCRIPTION:
Total 36 normal healthy adult male subjects will be enrolled in the study. Subjects will be administered either the Test or the Reference Product with 240 mL of water in each period as per the randomization schedule. Subjects will fast for at least 10 hours prior to dose administration and for at least 4 hours post dose. Standardized meals will be provided in each study period. Water will not be accessible to the subjects 1 hour Predose and 2 hours Post dose in each period. A total of 23 blood samples will be withdrawn for pharmacokinetic profiling. The whole blood concentrations of Tacrolimus will be measured by a validated LC/MS/MS analytical method. Ratio analysis will be performed for untransformed and log transformed pharmacokinetic parameters Cmax, AUC0-72, AUC0 inf. ANOVA will be performed on log transformed pharmacokinetic parameters Cmax, AUC0-72, AUC0-inf and 90% confidence interval will be constructed for the ratio of geometric least square mean of the Test and Reference products, obtained from the log-transformed data. Bioequivalence will be concluded if the ratio estimate as well as its 90% confidence interval, both falls within the acceptable range of 80.00% to 125.00% for Cmax, AUC0-72 and AUC0-inf.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects in the range of age from 18 to 55 years.
2. Body weight within ± 15% of ideal weight as related to height and body frame according to Life Insurance Corporation (LIC) Chart. (Appendix A)
3. Subjects with normal findings as determined by baseline history, physical examination and vital signs (blood pressure, pulse rate, respiration rate and axillary temperature).
4. Subjects with normal findings as determined by Haemogram with ESR, Biochemistry,Infectious Disease Screening (HIV, Hepatitis B and Hepatitis C) and Urinalysis, ECG, X-ray (X-ray if taken).
5. Willingness to follow the protocol requirement as evidenced by written, informed consent.
6. Agreeing to, not using any medication prescription and over the counter medications including vitamins and minerals for 14 days prior to study & during the course of the study.
7. No history or presence of significant alcoholism or drug abuse in the past one year.
8. Non-smokers, ex smokers and moderate smokers will be included. "Moderate smokers are defined as someone smoking 10 cigarettes or less per day, ex smokers are someone who completely stopped smoking for at least 3 months."

Exclusion Criteria:

1. Requiring medication for any ailment including enzyme-modifying drugs in the previous 28 days, before day 1 of dosing.
2. Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
3. History or presence of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic, haematological, gastrointestinal, endocrine, immunological or psychiatric diseases.
4. Participation in a clinical drug study or bioequivalence study 90 days prior to present study.
5. History or presence of malignancy or other serious diseases.
6. Refusal to abstain from food for at least ten (10) hours prior to administration of the study drug and for four (4) additional hours each, post dose during each study period.
7. Any contraindication to blood sampling.
8. Refusal to abstain from water for at least one (1) hour prior to study drug administration on dosing day of each study period and for at least two (2) additional hours, post dosing except 240 mL administered during administration of the dose.
9. Use of xanthine-containing beverages or food and grapefruit or grapefruit products for 48 hours prior to each drug dose.
10. Blood donation 90 days prior to the commencement of the study.
11. Subjects with positive HIV tests, HBsAg or Hepatitis-C tests.
12. Subjects having contradiction or hypersensitivity to Tacrolimus or related group of drugs or any excipients of the products.
13. Refusal to abstain from smoking or consumption of tobacco products 24 hours before dosing until last sample collection of each period.
14. Found positive in Breath alcohol test done at the time of screening or on the day of enrollment for each study period or for every ambulatory sample.
15. History or presence of problem in swallowing tablets or capsules.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-09; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To demonstrate bioequivalence between Test Product (A): Tacrolimus Capsules 1 mg manufactured by Panacea Biotec Limited, India and the corresponding Reference Product (B): Prograf (Tacrolimus) Capsules 1 mg manufactured by Astellas Pharma, Inc., USA | up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Suhas Khandave, Principal Investigator — Accutest Research Laboratories (I) Pvt. Ltd.
Locations (1):
- Accutest Research Laboratories (I) Pvt. Ltd., Navi Mumbai, Maharashtra, India